CLINICAL TRIAL: NCT03189459
Title: Reaching the Most Vulnerable: A Novel Model of Care in Advanced Parkinson's Disease
Brief Title: In-Home Care for Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17080209; 3994097 (Other Grant/Funding Number: NIH-NINDS)
Record Dates: First submitted 2017-05-25; First posted 2017-06-16 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: prospective cohort study (Aims 1 & 2) stepped wedge trial of caregiver peer mentoring (Aim 3)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HVP Patient-Subject (Active Comparator): Patients will be asked to participate in four study visits, which will involve in-home clinical assessments, a needs assessment, and completion of some questionnaires. Additional information will be obtained from patients' routine medical records: their medical and medication history, family history, neurological examination findings, and office visit records.
  Completion of Home Visit Program intervention.
  Interventions: Behavioral: Home Visit Program
- HVP Caregiver-Subject (Active Comparator): Caregivers enrolling in the study will be asked to participate in the four home visits, which will involve in-home clinical assessments and completion of some questionnaires. After the first home visit, caregivers will be matched with a peer mentor, an individual who was a prior caregiver to someone with PD who is interested in sharing their knowledge, experience, and time to help improve the lives of current caregivers. Once a week, for a period of 4 months between home visits 2 and 3, caregivers will be asked to meet with their peer mentor, who will be trained to serve as a resource and listening ear, in addition to the medical team.
  Completion of Home Visit Program and Caregiver Mentorship Program interventions.
  Interventions: Behavioral: Home Visit Program; Behavioral: Caregiver Mentorship Program
- De-identified Control Subjects (No Intervention): Control subjects will be drawn from the National Parkinson Foundation Parkinson Outcomes Project (POP). Patient-caregiver dyads will be matched on patient gender, age, and HY stage.
- HVP Peer Mentors (Active Comparator): Peer mentors enrolled in this study would be asked to complete a five-hour mentor training program. During this training, caregivers will be asked to complete some questionnaires about their background and caregiving experience. After completion of the mentorship training, peer mentors will be paired with a mentee who is a current caregiver enrolled in the home visit study along with their loved one with Parkinson's. Peer mentors will be asked to speak with their mentee once a week for 16 weeks. After a 16 week break, peer mentors will be paired with a second mentee and will repeat the process for another 16-week-long mentoring session.
  Completion of Caregiver Mentorship Program intervention.
  Interventions: Behavioral: Caregiver Mentorship Program

INTERVENTIONS:
Behavioral: Home Visit Program — RC: Informed consent discussion, documentation RN: UPDRS I-II, vitals, medication reconciliation, patient medical history and comorbidities RN and SW: Home safety assessment SW: Psychosocial assessment of dyad, HADS, assessment of mobility and homebound status, needs assessment of dyad, caregiver medical history and comorbidities RC: patient and caregiver short MoCA, PD-Rx, health literacy assessment, satisfaction surveys; patient PDQ-39/PDQ-8
  Arms: HVP Caregiver-Subject; HVP Patient-Subject
Behavioral: Caregiver Mentorship Program — Both mentors and mentees will be completing this program:
  Mentors will be asked to complete: 1) a Mentor Training - One 5-hour session at Rush University Medical Center; and 2) two 16-week periods of mentoring someone who is currently a caregiver for a patient with Parkinson's Disease
  Caregivers mentees will be asked to complete a 16 week mentorship program with their assigned mentor
  Arms: HVP Caregiver-Subject; HVP Peer Mentors

SUMMARY:
Advanced Parkinson's Disease is a debilitating, costly, and understudied condition. Improving access to comprehensive, specialized, in-home patient care and caregiver support offers the potential to minimize the downward spiral of morbidity and preventable healthcare utilization. The aim of this study is to test whether and to what degree an interdisciplinary home visit program, with and without peer mentoring for caregivers, will improve patient- and caregiver-reported outcomes and reduce healthcare costs when compared with usual care in advanced Parkinson's Disease.

DETAILED DESCRIPTION:
This interdisciplinary home visit program consists of 4 visits to patients' homes over the course of one year from a team of a movement disorders doctor, a nurse, a research coordinator, and a social worker. The team will come to a patient's home and assess the needs of both the patient and caregiver, and connect the patient with any needed services. These visits can replace or be in addition to seeing another movement disorders doctor.

As part of this study, not only would the patient receive home visits, but his/her caregiver would be paired with another caregiver from the community with lots of experience caring for someone with PD whose loved one may have passed away, but who volunteers to serve as a mentor. Current caregivers who enroll in the study will be asked to speak to their mentor once a week over a course of 4 months. These meetings can take place in person, by phone, or through video chat on an iPad that will be provided by our study team.

The information collected from the study participants will be compared to data available in the National Parkinson's Foundation's Parkinson's Outcome Project. The data will be matched according to age, gender, and disease severity.

ELIGIBILITY:
Inclusion Criteria:

HVP Patient-Subject

* Each subject must be 40 years of age or older. A subject may be of either gender, any race, and any ethnicity.
* Subjects must have a diagnosis of idiopathic Parkinson's Disease (inclusive of Parkinson's Disease Dementia) by a neurologist.
* Subjects will have been seen at least once in the past two years in the outpatient movement disorders clinic at Rush University Medical Center
* Subjects must be rated as HY stage 3-5 at the time of screening via chart review of the most recent clinical visit.
* Subjects must reside within a 60-minute public transit or driving distance of Rush University.
* Subjects must live at home (as defined by an independent dwelling such as an apartment, condominium, or house owned or rented by, or provided to/shared with the subject).
* Subjects must be home-bound according to the Medicare definition: "Leaving your home isn't recommended because of your condition; your condition keeps you from leaving home without help (such as using a wheelchair or walker, needing special transportation, or getting help from another person); leaving home takes a considerable and taxing effort." (http://www.medicare.gov/pubs/pdf/10969.pdf)
* Subjects have one or more of the following criteria, as determined by the referring neurologist: motor or cognitive fluctuations, multi-morbidity, medication mismanagement, cognitive impairment, symptoms of depression and/or anxiety, high risk for hospitalization or hospital readmission, high risk for nursing facility admission, suspected elder abuse, recent history of increased falls in home, caregiver burnout suspected, >2 cancelled or no-show appointments with the movement disorders providers in the preceding 12 months
* Subjects must have a caregiver willing to participate in the study, as defined by an unpaid individual cohabiting with or spending an average of >20 hours weekly engaged in care-related tasks related to the subject
* Subjects must either: 1) demonstrate capacity to consent, or 2) pending caregiver capacity assessment and caregiver consent, give assent or not dissent. Excluding individuals with cognitive impairment, dementia, depression, or psychosis would limit the generalizability of this study given the prevalence of each in advanced PD.

HVP Caregiver-Subject

* Each subject must be 30 years of age or older. A subject may be of either gender, any race, and any ethnicity.
* Each subject must be an unpaid individual cohabiting with or spending an average of >20 hours weekly engaged in care-related tasks related to the patient-subject. The caregiver-subject does not need to be the patient-subject's health care proxy or guardian.
* Each subject must demonstrate capacity to consent.
* Each subject must agree to participation in the nested trial of caregiver peer mentoring as a caregiver mentee
* Each subject must have a working telephone number at which he or she can be reached for check-in calls by the study team throughout the study.

Caregiver Peer Mentor

* Each subject must be 30 years of age or older. A subject may be of either gender, any race, and any ethnicity.
* Each subject must have >2 years of informal caregiving experience for an individual with PD or a related disorder.
* Each subject must have previously participated in a caregiver support group for PD, participated in a PD educational or outreach event, or given permission to be contacted for research.
* Each subject must be primarily English-speaking.
* Each subject must be willing and able to attend a one-time, five-hour mentor training session at Rush University
* Each subject must commit to two, 16-week blocks of peer mentoring either in person, by telephone, or by video conference on a study-provided iPad, for a minimum of 30 minutes weekly.
* Each subject must have a working telephone number at which he or she can be reached for check-in calls by the study team throughout the study.
* Each subject must be willing and able to attend a monthly, 45-minute supervision group during the two 16-week blocks of peer mentoring, held at Rush University.

De-identified Control Subjects

* Each subject must be 40 years of age or older. A subject may be of either gender, any race, and any ethnicity.
* Each subject must be a community-dwelling individual with idiopathic PD as diagnosed by a neurologist
* Each subject must be enrolled in the NPF POP at a US site.
* Each subject must have >2 consecutive, annual visits documented within the POP at which the subject is staged as HY 3-5.
* Each subject must have a caregiver participating in the POP at the above visits, as defined by completion of the MCSI.

Exclusion Criteria:

* Subjects exhibiting symptoms of a severe psychiatric disorder interfering with their ability to participate in the study, as determined by the referring neurologist, study team member, or PI.
* Subjects who are primarily non-English-speaking.

Exclusion Criteria for Subjects, by type:

HVP Patient-Subject

* Subjects with diagnoses of atypical parkinsonism or possible/probable PSP, MSA, CBS,or DLB will be excluded.
* Subjects without an informal caregiver will be excluded.

HVP Caregiver-Subject

* Active psychosis or other severe psychiatric disease
* Terminal illness (life expectancy <12 months)

Caregiver Peer Mentor

* Active psychosis or other severe psychiatric disease
* Terminal illness (life expectancy <12 months)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Quality of Life using the PDQ-39 | 1 year
  Assesses Parkinson's disease-specific health related quality before and after participation in the home visit program

SECONDARY OUTCOMES:
Caregiver Strain using the MCSI | 1 year
  Assesses caregiver strain over the course of the home visit program
Effectiveness of Peer Mentoring using the HADS | 16 weeks
  Assesses the anxiety and depression of mentees and mentors before and after participation in the mentorship program

CONTACTS AND LOCATIONS:
Overall Officials: Jori Fleisher, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Fleisher JE, Suresh M, Klostermann EC, Lee J, Hess SP, Myrick E, Mitchem D, Woo K, Sennott BJ, Witek NP, Chen SM, Beck JC, Ouyang B, Wilkinson JR, Hall DA, Chodosh J. IN-HOME-PDCaregivers: The effects of a combined home visit and peer mentoring intervention for caregivers of homebound individuals with advanced Parkinson's disease. Parkinsonism Relat Disord. 2023 Jan;106:105222. doi: 10.1016/j.parkreldis.2022.11.014. Epub 2022 Nov 17. PMID 36446676
- [Derived] Fleisher JE, Hess SP, Klostermann EC, Lee J, Myrick E, Mitchem D, Niemet C, Woo K, Sennott BJ, Sanghvi M, Witek N, Beck JC, Wilkinson JR, Ouyang B, Hall DA, Chodosh J. IN-HOME-PD: The effects of longitudinal telehealth-enhanced interdisciplinary home visits on care and quality of life for homebound individuals with Parkinson's disease. Parkinsonism Relat Disord. 2022 Sep;102:68-76. doi: 10.1016/j.parkreldis.2022.07.017. Epub 2022 Aug 7. PMID 35963046
- [Derived] Fleisher JE, Akram F, Lee J, Klostermann EC, Hess SP, Myrick E, Levin M, Ouyang B, Wilkinson J, Hall DA, Chodosh J. Peer Mentoring Program for Informal Caregivers of Homebound Individuals With Advanced Parkinson Disease (Share the Care): Protocol for a Single-Center, Crossover Pilot Study. JMIR Res Protoc. 2022 May 26;11(5):e34750. doi: 10.2196/34750. PMID 35481819
- [Derived] Fleisher JE, Hess S, Sennott BJ, Myrick E, Wallace EK, Lee J, Sanghvi M, Woo K, Ouyang B, Wilkinson JR, Beck J, Johnson TJ, Hall DA, Chodosh J. Longitudinal, Interdisciplinary Home Visits Versus Usual Care for Homebound People With Advanced Parkinson Disease: Protocol for a Controlled Trial. JMIR Res Protoc. 2021 Sep 14;10(9):e31690. doi: 10.2196/31690. PMID 34238753

DOCUMENTS (3):
  • Informed Consent Form: _CaregiverPeerMentor (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03189459/ICF_000.pdf
  • Informed Consent Form: _Caregiver (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03189459/ICF_001.pdf
  • Informed Consent Form: _Patient (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03189459/ICF_002.pdf